CLINICAL TRIAL: NCT06526026
Title: An Innovative Mental Health Virtual Ward: Evaluation of Patient-Centered Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS26297
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Disorder; Mental Health Impairment; Psychiatric Emergency; Crisis; Emotional
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Health Virtual Ward (Experimental): Admission to the Mental Health Virtual Ward
  Interventions: Behavioral: Virtual crisis stabilization support with a multi-disciplinary team

INTERVENTIONS:
Behavioral: Virtual crisis stabilization support with a multi-disciplinary team — Daily 1:1 sessions with multidisciplinary team via a range of virtual modalities (videoconferencing, phone, text, email), group programming, self-management resources, remote home monitoring app, referrals and linkages to community programs.

SUMMARY:
The goal of this study is to evaluate if admission to the Mental Health Virtual Ward (MH vWard) for mental health crisis stabilization is having a meaningful positive impact on patient reported outcomes and healthcare utilization. The objectives of this study are:

1. Prospectively measure demographic, recovery, service delivery, and systems use outcomes in a cohort of MH vWard admissions.
2. establish this cohort for use in future research.

As part of the intervention, participants will receive care in the MH vWard for an average of 5 days following a visit to an emergency department or crisis centre for a mental health crisis. While admitted to the MH vWard, participants will:

1. Engage in individual therapy and care planning with a clinician or psychiatry team.
2. Have engagement with formal (community providers) and informal supports (family, friends) for collateral and collaboration.
3. Receive medication reconciliation and management.
4. Participate in group programming.
5. Receive referrals for follow-up services.
6. Have access to after hours support.
7. Have access to the Telus Home Health Monitoring (HHM) App, which is custom designed to complement the services provided by the program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals admitted to the Mental Health Virtual Ward.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
The World Health Organization-Five (WHO-5) Well-Being Index | 1 week, 5 weeks and 6 months from date of discharge
  The World Health Organization-Five (WHO-5) Well-Being Index is a questionnaire used for the assessment of subjective psychological well-being.
  Five questions are answered on a scale of 1-5 (0 meaning the individual agrees with the statement "at no time", 5 meaning they agree with the statement "all of the time").
  Minimum value: 0 Maximum value: 25 A higher score represents better quality of life and well-being, a lower score represents lower quality of life and well-being.

SECONDARY OUTCOMES:
Post-discharge Healthcare Utilization (self-report) | 1 week post discharge, 5 weeks post discharge and 6 months from date of discharge
  Number of participants who self-report further healthcare utilization following discharge from the virtual ward (all participants)
  Systems use outcomes will include: emergency department visits, crisis centre visits, and psychiatric hospitalizations collected by self-report. Patients can answer questionnaires electronically, over the phone, or in person with a member of the research team.
Post-discharge Healthcare Utilization (administrative data) | 1 week post discharge, 5 weeks post discharge and 6 months from date of discharge
  Number of participants with administrative data supporting further healthcare utilization following discharge from the virtual ward (urban participants only)
  Systems use outcomes will include: emergency department visits, crisis centre visits, and psychiatric hospitalizations collected via healthcare administrative data. This data will be used to collect some systems use outcomes data on participants lost to follow-up in the study, as well as allow for the assessment of recall bias when compared to self-reporting of healthcare utilization.
Maryland Assessment of Recovery Scale-Twelve (MARS-12) | 1 week post discharge, 5 weeks post discharge, 6 months post-discharge
  Maryland Assessment of Recovery Scale-Twelve (MARS-12) contains a list of statements about an individuals subjective attitude and beliefs towards their own health an wellness.
  Twelve questions are answered on a scale from 1-5 (1 meaning the participant "not at all" agrees with the statement, 5 meaning the participant "very much" agrees with the statement).
  Minimum value: 12 Maximum value: 60 A higher score represents a higher personal recovery post-discharge, a lower score represent a lower personal recovery post-discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hensel, MD, Principal Investigator — University of Manitoba and Shared Health Manitoba/Psychiatry
Locations (1):
- Crisis Stabilization Unit, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo BA, Shterenberg R, Bolton JM, Dewa CS, Pullia K, Hensel JM. Virtual Acute Psychiatric Ward: Evaluation of Outcomes and Cost Savings. Psychiatr Serv. 2023 Oct 1;74(10):1045-1051. doi: 10.1176/appi.ps.20220332. Epub 2023 Apr 5. PMID 37016824
- [Background] Pullia K, Clavio A, Bolton JM, Hunzinger E, Svenne S, Hensel JM. Providing crisis care in a pandemic: a virtual based crisis stabilization unit. Front Health Serv. 2023 May 16;3:1030396. doi: 10.3389/frhs.2023.1030396. eCollection 2023. PMID 37260632
- [Background] Palay J, Taillieu TL, Afifi TO, Turner S, Bolton JM, Enns MW, Smith M, Lesage A, Bakal JA, Rush B, Adair CE, Vigod SN, Clelland S, Rittenbach K, Kurdyak P, Sareen J. Prevalence of Mental Disorders and Suicidality in Canadian Provinces. Can J Psychiatry. 2019 Nov;64(11):761-769. doi: 10.1177/0706743719878987. Epub 2019 Oct 16. PMID 31619055
- [Background] Butler A, Adair C, Jones W, et al. Towards quality mental health services in Canada: a comparison of performance indicators across 5 provinces. Vancouver, BC: Centre for Applied
- [Background] Shared Health (2018). Shared Health Mental Health Program STATs 2018.
- [Background] Crisis Response Services (2022). Crisis Response Services Annual Performance Report April 1, 2021-Mrach 31, 2022
- [Background] Canadian Institute for Health Information, 2016.
- [Background] Hensel JM, Bolton JM, Svenne DC, Ulrich L. Innovation through virtualization: Crisis mental health care during Covid-19. Canadian Journal of Community Mental Health. 2020 Nov 2;39(2):71-5.
- [Background] Arsenault-Lapierre G, Henein M, Gaid D, Le Berre M, Gore G, Vedel I. Hospital-at-Home Interventions vs In-Hospital Stay for Patients With Chronic Disease Who Present to the Emergency Department: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Jun 1;4(6):e2111568. doi: 10.1001/jamanetworkopen.2021.11568. PMID 34100939
- [Background] Lee K, Bolton SL, Shterenberg R, Bolton JM, Hensel JM. Early Learning From a Low-Resource COVID-Response Virtual Mental Health Crisis Ward: Mixed Methods Study. JMIR Form Res. 2022 Nov 4;6(11):e39861. doi: 10.2196/39861. PMID 36252139
- [Background] Ramsay C, Pickard R, Robertson C, Close A, Vale L, Armstrong N, Barocas DA, Eden CG, Fraser C, Gurung T, Jenkinson D, Jia X, Lam TB, Mowatt G, Neal DE, Robinson MC, Royle J, Rushton SP, Sharma P, Shirley MD, Soomro N. Systematic review and economic modelling of the relative clinical benefit and cost-effectiveness of laparoscopic surgery and robotic surgery for removal of the prostate in men with localised prostate cancer. Health Technol Assess. 2012;16(41):1-313. doi: 10.3310/hta16410. PMID 23127367
- [Background] Frank L, Basch E, Selby JV; Patient-Centered Outcomes Research Institute. The PCORI perspective on patient-centered outcomes research. JAMA. 2014 Oct 15;312(15):1513-4. doi: 10.1001/jama.2014.11100. No abstract available. PMID 25167382
- [Background] Bhattacharyya O, Hayden L, Hensel J. Health Services and Designing for Uncertainty: How a "lean startup" approach can help create an effective community-based program. Stanford Social Innovation Review. 2015;doi:10.48558/kw2z-6a08
- [Background] Computerised cognitive behaviour therapy (cCBT) as treatment for depression in primary care (REEACT trial): large scale pragmatic randomised controlled trial. BMJ. 2016 Jan 12;352:i195. doi: 10.1136/bmj.i195. No abstract available. PMID 26759375
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Newnham EA, Hooke GR, Page AC. Monitoring treatment response and outcomes using the World Health Organization's Wellbeing Index in psychiatric care. J Affect Disord. 2010 Apr;122(1-2):133-8. doi: 10.1016/j.jad.2009.06.005. Epub 2009 Jul 9. PMID 19592116
- [Background] Idiculla T, Eisen S. Integrating science and practice. The BASIS-24 Behavior and symptom identification scale. ResearchGate. 2012; 2(2):16-19.
- [Background] Eisen SV, Normand SL, Belanger AJ, Spiro A 3rd, Esch D. The Revised Behavior and Symptom Identification Scale (BASIS-R): reliability and validity. Med Care. 2004 Dec;42(12):1230-41. doi: 10.1097/00005650-200412000-00010. PMID 15550803
- [Background] Drapalski AL, Medoff D, Unick GJ, Velligan DI, Dixon LB, Bellack AS. Assessing recovery of people with serious mental illness: development of a new scale. Psychiatr Serv. 2012 Jan;63(1):48-53. doi: 10.1176/appi.ps.201100109. PMID 22227759

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT06526026/Prot_SAP_001.pdf